CLINICAL TRIAL: NCT00664196
Title: Phase Ia/Ib Trial of Anti-PSMA Designer T Cells in Advanced Prostate Cancer After Non-Myeloablative Conditioning
Brief Title: Trial of Anti-PSMA Designer T Cells in Advanced Prostate Cancer After Non-Myeloablative Conditioning
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 595-04; W81XWH-05-1-0408
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; T cells; Gene Transfer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Gene Modified T Cells

INTERVENTIONS:
Biological: Gene Modified T Cells — One time infusion Modified T-Cells given through a vein in the arm or a catheter over a 30-60 minute period.
  Other Names: Designer T-Cells; PSMA; Hormone Refractory

SUMMARY:
This study tests the safety and tolerability of autologous anti-PSMA gene-modified T cells (designer T cells) in hormone refractory prostate cancer.

DETAILED DESCRIPTION:
The study creates autologous gene-modified T cells against prostate specific membrane antigen (PSMA, unrelated to PSA) (designer T cells) by ex vivo modification of patient T cells. T cells are collected by leukopheresis, transported to the RWMC cGMP Cell Manipulation Core and transduced with retrovirus containing a chimeric antigen receptor (CAR) that is expressed on the modified cells. This CAR links specificity of an antibody against PSMA with signaling domains of the T cell and redirects the recognition of the T cells to engage and kill prostate cancer cells anywhere in the body. These are administered at a dose of 10^10 with randomization to either low or moderate Interleukin 2 given by CI (continuous infusion) for one month following the T cell infusion. Subsequent subjects will receive 10^11 cells with Interleukin 2 at either low or moderate dose, in a non randomized manner, depending upon the outcome of the prior cohort. Prior to T cell infusion, all subjects will receive non-myeloablative (NMA) conditioning. This conditioning creates a "space" in the blood and marrow for engraftment of the infused cells to maintain of high level of anti-tumor effector T cells in the body. Each patient is treated with a single dose of T cells, without repeat dosing. Patients are followed for toxicity and response and pharmacokinetics-pharmacodynamics of the infused T cells. Patients are on-study for one-month after their T cell dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of prostate cancer
2. Elevated PSA
3. Life expectancy > 4 months
4. Performance status 0-1
5. ANC 1.0
6. Platelets > 100,000
7. Hemoglobin > 8.0
8. Creatinine < 1.5mg/dl
9. Direct Bilirubin < 1.5 mg/dl
10. No evidence of CHF, CAD, cardiac arrhythmias, A-fib, A flutter, myocardial infarction.
11. No serious, symptomatic obstructive or emphysematous lung disease
12. No asthma requiring IV medication during last 12 months, no serious lung disease associated with dyspnea at normal activity levels, or at rest due to any cause, including cancer metastasis and pleural effusion
13. Patients must have a biopsy able tumor, and be willing to undergo biopsy (Group 3 only)
14. Patient is at least 18 years of age.

Exclusion Criteria:

1. Serious or unstable renal, hepatic, pulmonary, cardiovascular, endocrine, rheumatologic or allergic disease based on history, labs or physical exam
2. Active clinical disease caused by CMV, Hepatitis B, or C, HIV, TB
3. Cytotoxic and/or radiation therapy during last 4 weeks prior to entry
4. Any concurrent malignancies
5. Patient requires systemic steroids
6. Patient has participated in prior investigational therapy
7. Patient has prior exposure to mouse antibody
8. Patient has had irradiation to whole pelvis or >25% marrow

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of using modified T cells by documenting the type and severity of any side effects and establishing the Maximum Tolerated Dose (MTD) | 1 Month

SECONDARY OUTCOMES:
Tumor Response | 1 Month
Pharmacokinetics | 1 Month
Pharmacodynamics | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Junghans, PhD, MD, Principal Investigator — Roger Williams Hospital
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States